CLINICAL TRIAL: NCT06843525
Title: Exploring a Neuropathic Basis for Acute Pulpal Pain- a Clinical Pilot
Brief Title: Bite Force Measurements
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: New Jersey Alliance for Clinical and Translational Science (Unknown)
Responsible Party: Principal Investigator, Gayathri Subramanian, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2024002660
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Irreversible Pulpitis; Apical Periodontitis; Pulpal Necrosis
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Controls: Patients who require a restoration on a vital but carious lower 1st or second molar tooth
- Affected Pulp/Healthy Apex: Patients who have a carious 1st or second lower molar tooth with pulpal involvement in a vital tooth
- Diseased Pulp/ Healthy Apex: Patients who experience irreversible pulpitis or pulpal necrosis in a lower 1st or second molar tooth
- Diseased Pulp/Diseased Apex: Patients who experience irreversible pulpitis or pulpal necrosis in a lower 1st or second molar tooth and have tenderness to palpation/percussion due to apical periodontitis or demonstrate radiographic evidence of periapical pathology

SUMMARY:
ABSTRACT: Acute dental pain from untreated decay often drives patients to emergency rooms (ERs), where the lack of definitive dental treatment results in nearly 75% of these patients receiving analgesics, predominantly opioids. Addressing the need for non-opioid pain alternatives is crucial. Emerging evidence suggests that dental pain from pulpal and periodontal conditions (affecting the tooth's nerve and surrounding tissues) involves neuropathic mechanisms, such as mechanical allodynia (MA) and central sensitization (CS). These mechanisms can amplify pain perception, causing typically non-painful actions, like chewing, to become painful and resulting in hypersensitivity extending beyond the affected tooth. Reliably identifying these mechanisms with quantitative measures can support improved pain assessment and targeted non-opioid treatment. This minimally invasive prospective cohort study will use the FDA-approved Innobyte® device, a precise bite-force measurement tool, to evaluate periodontal health and to quantify mechanical pain thresholds in patients requiring endodontic treatment (root canal therapy).

DETAILED DESCRIPTION:
This study aims to validate neuropathic mechanisms as therapeutic targets by quantifying toothache-induced mechanical allodynia. It could potentially support the use of neuropathic pain medications, like gabapentin, as adjuncts to traditional pain management. The study's findings could also reduce opioid reliance in ER settings, particularly benefiting underserved populations with limited access to dental care. This innovative approach challenges conventional views on dental pain and may provide the foundation for future research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who present for
* a lower 1st or 2nd molar filling in an otherwise healthy tooth, i.e., does not have large decay that has already infected the nerve of the tooth, or there is increased mobility due to gum disease or a root canal treatment on a lower molar tooth and there is no history of injury to the tooth, or
* a lower molar root canal treatment, and
* are 18 years or older
* capable of providing informed consent, are eligible to participate in the study, as long as they satisfy the criteria below.
* The opposing tooth is present, symptom-free and has adequate tooth structure that allows it to make contact with the tooth it bites against, and
* are English-speaking

Exclusion Criteria:

* Any patient, even if satisfying the criteria above, may not take part if any of the below is true:
* Compromised ability to guard their self-interest, for e.g., prisoners, children, pregnant women, patients with intellectual/cognitive disability are not enrolled in the study.
* Take prescription pain medications for long-standing health conditions
* Addiction/ substance dependence
* Swelling that extends beyond the tooth in question
* Are already taking an antibiotic to treat an infection/swelling
* Missing complementary molar on the same or opposite side of the mouth
* Missing more than 2 teeth in a quadrant (other than 3rd molars)
* Any other molar in the pair either on the side of the tooth of interest or the molar pair on the other side is painful to biting pressure or upon 'tapping' the tooth with the handle of the mouth mirror
* The patient has taken a pain medication within the last 6 hours

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who present to Rutgers School of Dental Medicine for a lower 1st or 2nd molar filling in an otherwise healthy tooth, i.e., does not have large decay that has already infected the nerve of the tooth, or there is increased mobility due to gum disease or a root canal treatment on a lower molar tooth and there is no history of injury to the tooth, or for a lower molar root canal treatment in the 1st or second molar tooth will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical Allodynia | Baseline
  Ipsilateral full arch and tooth specific bite-force
Mechanical Allodynia | 10 minutes post-local anesthesia
  Ipsilateral full arch and tooth specific bite-force
Central Sensitization | Baseline
  Contralateral tooth specific bite-force
Central Sensitization | 10 minutes post-local anesthesia
  Contralateral tooth specific bite-force

SECONDARY OUTCOMES:
Assessment of tooth vitality | Baseline
  Cold Test and Electric Pulp Test
Assessment of tooth vitality | 10 minutes post-local anesthesia
  Cold Test and Electric Pulp Test
Numerical Pain Rating Score | Baseline
  Patient-reported pain on 0-10 scale
Numerical Pain Rating Score | 10 minutes post-local anesthesia
  Patient-reported pain on 0-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Varvara Vanessa Chrepa, DDS, MS, PhD, Principal Investigator — Rutgers School of Dental Medicine; Gayathri Subramanian, PhD, DMD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the key results of the study will be available after deidentification to individuals submitting a written request. The study protocol and informed consent documents, and aggregate data will be shared on ClinicalTrials.gov. The data will be made available about 9 months and ending 36 months after publication, if the investigators whose proposed use of the data has been approved by an independent review committee.
Supporting Information: Study Protocol, ICF
Time Frame: A year after completion of the study and data analysis
Access Criteria: Individual participant data that underlie the key results of the study will be available after deidentification to individuals submitting a written request. The study protocol and informed consent documents, and aggregate data will be shared on ClinicalTrials.gov. The data will be made available about 9 months and ending 36 months after publication, if the investigators whose proposed use of the data has been approved by an independent review committee.